CLINICAL TRIAL: NCT05292703
Title: Olfaction, Virtual Reality and Art in Health
Acronym: OREVAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-PP-01
Record Dates: First submitted 2022-03-01; First posted 2022-03-23 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Elderly People

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- face-to-face group (Experimental): In the face-to-face group, the intervention is a participatory activity based on art and olfactory stimulation which consists of practicing art in a group under supervision, involving the participants directly in the creative process, allowing them to become co-authors. Participants will meet once a week for 4 weeks for a 2-hour workshop at the Institut Claude Pompidou in Nice in a dedicated space, adapted to health circumstances and respecting social distancing measures. Due to the health crisis, the workshops will be offered in several groups ranging from 8 to 10 participants, these groups will be equal. A different theme will be offered each week. Each workshop will be led by the same artist who will propose creative activities to be carried out by the participants and each session will result in a creation that the participant will take away, bringing into play artistic skills and olfactory identification capacities
  Interventions: Other: Participatory activity based on art and olfactory stimulation
- remote group (Experimental): For the remote group, immediately after randomization, they will receive the connection link to the internet application and an individual connection code. The intervention is a participative activity based on art and olfactory stimulation which consists of practicing art virtually in conjunction with olfactory identification by following a dedicated program developed in partnership with the same artist involved in the workshops in presence, so that the virtual activities are very similar to those of the face-to-face workshop. The artistic workshops will take place according to 4 themes with a different theme per week. Each workshop end with an original artistic creation received by email, bringing into play artistic skills and olfactory identification capacities. Each participant will connect once a week at their convenience during 4 weeks.
  Interventions: Other: practicing art virtually in conjunction with olfactory identification

INTERVENTIONS:
Other: Participatory activity based on art and olfactory stimulation — practicing art in a group under supervision, involving the participants directly in the creative process, allowing them to become co-authors. Participants will meet once a week for 4 weeks for a 2-hour workshop at the Institut Claude Pompidou in Nice in a dedicated space, A different theme will be offered each week. Each workshop will be led by the same artist who will propose creative activities to be carried out by the participants and each session will result in a creation that the participant will take away, bringing into play artistic skills and olfactory identification capacities.
  Arms: face-to-face group
Other: practicing art virtually in conjunction with olfactory identification — For the remote group, , they will receive the connection link to the internet application and an individual connection code.
  The intervention is a participative activity based on art and olfactory stimulation which consists of practicing art virtually in conjunction with olfactory identification by following a dedicated program developed in partnership with the same artist involved in the workshops in presence, so that the virtual activities are very similar to those of the face-to-face workshop.
  The artistic workshops will take place according to 4 themes with a different theme per week. Each workshop end with an original artistic creation received by email, bringing into play artistic skills and olfactory identification capacities. Each participant will connect once a week at their convenience during 4 weeks.
  Arms: remote group

SUMMARY:
The main objective of this study is to compare the well-being of a group of seniors participating for a month in face-to-face sessions of artistic and olfactory activities with another group of seniors performing the same type of activity for a month but remotely with connection to a dedicated application.

Well-being, Quality of Life, Health, Apathy and Olfactory identification scales are proposed before the intervention, at the end of the intervention (V0, V1), then 3 months after the end of the intervention. A Usability Evaluation questionnaire will be sent to the participants of the remote group after use (V1).

DETAILED DESCRIPTION:
Health is defined by WHO as a condition of mental, physical and social well-being. Cognitive aging markers have been defined such as apathy and deterioration of olfactory identification. Artistic creation can be used to improve health, and olfactory stimulation can improve olfactory abilities.

The main objective of this study is to compare the well-being of a group of seniors participating for a month in face-to-face sessions of artistic and olfactory activities with another group of seniors performing the same type of activity for a month but remotely with connection to a dedicated application.

Well-being, Quality of Life, Health, Apathy and Olfactory identification scales are proposed before the intervention, at the end of the intervention (V0, V1), then 3 months after the end of the intervention. A Usability Evaluation questionnaire will be sent to the participants of the remote group after use (V1).

Concerning the categorical variables, the frequencies will be calculated. First the basic characteristics (age, sex, etc.) will be described and compared for each group (i.e., intervention versus control) using parametric and non-parametric tests according to the distribution of variables. Regarding the quantitative variables, the distribution will be studied (mean, median, mode, minimum, maximum, confidence interval around the mean, standard deviation). The statistical tests used will be unpaired T-tests or Mann-Whitney U-tests to compare the two appropriate groups depending on the groups.

Several effects are expected following the practice of participatory artistic workshops. First, an improvement in well-being is expected, measured by the WEMBS scale. An immediate and medium-term benefit is expected, which will be measured 3 months after the end of the workshops. In a second step, an improvement in the Quality of Life and the state of Health is expected. Measurement data for early markers of cognitive decline, Apathy and Olfactory identification should improve. In the long term and more generally, the validation of the proposed study could make it possible to legitimately ensure its dissemination on a larger scale, and to strengthen the involvement of seniors with public users in participatory artistic programs in person or remotely, in order to ensure them a quality ageing. The data will be compared a posteriori with international data in order to compare the effects of artistic workshops in person or remotely. An acceptability questionnaire will assess the adherence of seniors to a distance and virtual artistic program before and after use.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 or more
* Get internet access and an electronic tool such as a smartphone or tablet,
* Be fluent in French language.
* Be available during participatory artistic workshop sessions.
* Be affiliated with Social Security

Exclusion Criteria:

* Not fluent in french language,
* Present sensory and/or cognitive deterioration identified by the investigator during inclusion,
* Being under guardianship or curatorship or safeguard of justice,
* Being unable to give or sign consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
change in Warwick-Edinburgh Mental Well-Being Scale (WEMBS) | At the beginning, after the session and 3 months after the end of the session
  The 14-item scale WEMWBS has 5 response categories, summed to provide a single score. The items are all worded positively and cover both feeling and functioning aspects of mental wellbeing, thereby making the concept more accessible.

SECONDARY OUTCOMES:
Quality of life scale (EQ5D) | At the beginning, after the session and 3 months after the end of the session
  EQ-5D, ranking from 1 to 5, 1= no problems, 2= light, 2= moderate; 3= severe; 5= very severe
Health scale (CESAM) | At the beginning, after the session and 3 months after the end of the session
  CESAM provides two complementary information:
  1. A global score of frailty ranged from 0 (i.e., best health and functional condition) to 18 (i.e., worse health and functional condition) and
  2. Categorized health condition in four levels (vigorous with a score between 0 and 3, mild frailty with a score between 4 and 7, moderate frailty with a score between 8 and 12, and important frailty with a score above 12
Apathy scale (b-DAS) | At the beginning, after the session and 3 months after the end of the session
  Das-short: min 12-max 21, executive dimension: min 3- max 6, cut-off 4-5; emotional dimension min 4- max 7, cut-off 5-6; Initiation dimension min 5- max 8, cut-off 6-7
User experience evaluation questionnaire (Usability Evaluation) | After the session and 3 months after the end of the session
  satisfaction assessment
Olfactory identification test (Bellecôte) | At the beginning, after the session et 3 months after the end of the session
  rating from 0 to 6; normal identification >4

CONTACTS AND LOCATIONS:
Overall Officials: AURIANE GROS, SPEECH THERAPIST, Principal Investigator — CMRR
Locations (1):
- CHU de Nice Centre Mémoire, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided